CLINICAL TRIAL: NCT02883582
Title: Adjuvant Therapy for Severe Asthma by an Oxyhydrogen Generator With Nebulizer: A Multi-centric, Randomized, Parallel-control and Double-blinded Clinic Study on Effectiveness and Safety
Brief Title: Adjuvant Therapy for Severe Asthma by an Oxyhydrogen Generator With Nebulizer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Asclepius Meditec Inc. (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); The Second Hospital of Hebei Medical University (Other); Tianjin Medical University General Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLZhang
Record Dates: First submitted 2016-08-15; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: asthma ,hydrogen
MeSH Terms: conditions — Asthma | interventions — Nebulizers and Vaporizers; Oxygen Inhalation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxyhydrogen (Experimental): conventional treatment (bronchodilator (LABA,LAMA)with or without ICS)+ hydrogen/ oxygen inhaled
  Interventions: Device: oxyhydrogen
- oxygen (Experimental): conventional treatment (bronchodilator (LABA,LAMA) with or without ICS)+ oxygen inhaled
  Interventions: Device: oxygen

INTERVENTIONS:
Device: oxyhydrogen — Hydrogen/oxygen mixed gas inhaled(proportion 2:1),3 L/min . 1 hour each time,twice a day(BID).Test Duration is three months.
  Other Names: oxyhydrogen generator with nebulizer
  Arms: oxyhydrogen
Device: oxygen — oxygen inhaled,3 L/min . 1 hour each time,twice a day(BID).Test Duration is three months.
  Other Names: Medical molecular sieve oxygenerator
  Arms: oxygen

SUMMARY:
The purpose for the trial is intended to evaluate safety and effectiveness of an oxyhydrogen generator with nebulizer in an adjuvant therapy for patients with severe asthma.

DETAILED DESCRIPTION:
The oxyhydrogen generator with nebulizer in (treatment group) or control group was applied randomly for the patients with severe asthma in this study, then the therapeutic effects from both treatment and control groups were analyzed and evaluated to verify its safety and effectiveness.This study is a multi-center, randomized, double-blind study. Each patient was expected to participate in the trial for 104±3 day.The screening period was 14±1 days, and the subjects would continue to be applied with the previous asthma treatment scheme. The primary objective was to collect the baseline data related to the subjects.The patients would receive 30±1 day of treatment with the product; after that, observation of 60±1 days was required.Total patients number is 150 cases, of which 75 cases are treatment group and the others are control group.All cases respectively are distributed in 5 clinical hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: ≥18 years old but ≤65 years old; sex unlimited;
2. The subjects were required to be suffered with asthma for 6 months at least by clinical diagnosis by the respirologist based on the international standards (GINA2012).There was the support of one of the following objective evidences in screening and treatment or five years before the treatment:

   * It was the positive reaction in the methacholine provocative test (for the patients not applied with inhaled corticosteroid (ICS) were required at PC20<8mg/mL and PD20<0.7mg; for the patients applied with ICS were required at PC20<16mg/mL or PD20<1.4mg);

     * The airway reversibility test, with a positive reaction, was defined asΔFEV1.0% at a basis FEV1.0≥200mL at 30 minutes after 400μgsalbutamol aerosol (mist-storing bottle might be used deliberately) was inhaled; ③ The peak expiratory flow (PEF) aberration rate>20% (that is, the difference or average value of maximum and minimum PEFs times 100); it was measured for seven days successively;

       * The reaction record after asthma maintenance treatment for one course of treatment (e.g. four weeks) (defined as ΔFEV1.0 and its absolute value≥200mL);
3. According with severe asthma diagnosis: The drug therapy was required for Level-4 and 5 asthma according to GINA Guide in the past year (The large dose of ICS combined LABA or leukotriene modifier/theophyline), or the systemic corticosteroid treatment lasted at ≥50% of the time to prevent from the "uncontrollable" asthma; or the "uncontrollable" asthma still occurred even if in above treatment. The uncontrollable asthma should meet one of the following requirements at least:

   * Symptom control difference: ACQ>1.5, and ACT<20 (or "Non-good control" in GINA Guide);

     * Frequent severe attack: Receiving systemic corticosteroid treatment for more than twice in the past year (over three days each time); ③ Serious attack: Hospitalizing once in ICU or mechanical ventilation at least in the past year; ④ Airway limitation: After bronchodilator was stopped properly, FEVl.0%<80% (FEV/FVC decreased to be less than lower limit of the normal value). The controlled asthma deteriorated at the decrement of above large dose ICS or systemic corticosteroid (or combined biologic agent);
4. The subjects or their legal agents could understand the trial objectives, demonstrating the compliance to the trail scheme, and signed the Informed Consent Form.

Exclusion Criteria:

1. The subjects at a body mass index>38kg/m2, or a weight<40kg;
2. The subjects' smoking amount>10 packages times the year number (e.g. number of cigarettes × the number of years for smoking/20);
3. Based on clinical interview, experience or screening inspection results, the subjects should participate in this trial improperly if the doctor responsible for the trial believed there was risk when they participated in the trial, or the research results were affected;
4. The subjects who had the recreational drug abuse history or other allergic history, but the doctor responsible for the trial believed these subjects limited by the history could participated in the trial;
5. The women subjects who were in the pregnancy or suckling period, or six weeks at least after delivery, or stopped breastfeeding for six weeks. If the women subjects were found to be pregnant in receiving one inspection, then, the inspection data for this item should be rejected in analysis;
6. The subjects ever participated in the study on a new drug or any other drugs, and were within 3 months for the first administration, or every participated in one research involved in invasive operation within 3 months. Any research evaluation should be put off to three months later in the first administration or invasive operation when they participated in the research. It was approved by the steering committee if the subjects participating in other researches were included in trial groups or continued participating in this research;
7. The investigator believed the subjects showed the risk of non-compliance with research procedures;
8. The subjects had the mental disease history resulting in loss of active ability in the recent period;
9. The following disease history or evidences demonstrated within two weeks in baseline assessment that the subjects suffered upper or lower respiratory infections or related symptoms (including common cold) (the assessment should be put off);
10. The subject changed the asthmatic drugs within four weeks before the screening;
11. The subject suffered the asthma attack in the month prior (administered with systemic corticosteroid or temporarily increasing oral corticosteroid at three days of stable base dose at least);
12. Other important diagnoses possibly similar to asthma or complicated asthma, especially respiratory dysfunction, panic attack and evident social psychological problems (if these diagnoses were seen as the patient's main symptoms rather than the symptoms except severe asthma);
13. Other severe primary pulmonary diseases, especially pulmonary embolism, pulmonary hypertension, interstitial pulmonary disease and lung cancer;
14. The subjects with emphysema and bronchiectasis should be excluded only when these diagnoses are considered as their main symptoms rather than other symptoms except severe asthma;
15. The subjects who were diagnosed with other chronic inflammatory diseases (inflammatory bowel disease, rheumatoid arthritis) except asthma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
differentials from Mini Asthma Quality of life questionnaire (Mini AQLQ) | at 3 months
  Mini Asthma Quality of life questionnaire (Mini AQLQ) was used for evaluation on asthma treatment after the subjects were treated, to determine the product effectiveness.

SECONDARY OUTCOMES:
differentials from asthma control questionnaire | at 3 months
  the asthma control questionnaire (ACQ) was used for the evaluation on the subjects' asthma state after treatment, to determine effectiveness of the product.
differentials from asthma control test (ACT) | at 3 months
  The asthma control test (ACT) is used for evaluation of the asthma state after treatment, to determine effectiveness of the product.
differentials from Peak Expiratory Flow (PEF) daily aberration rate | at 3 months
  Peak Expiratory Flow (PEF) refers to the instant flow rate in the fastest expiratory flow in the forced vital capacity measurement process, mainly reflecting the strength of respiratory flow and airway obstruction.
differentials from airway resistance measurement | at 3 months
  The patient airway resistance was measured was measured, including: Rat5Hz, Rat20Hz, Xat5Hz, MeanR5~R20 and AX.
differentials from number of asthma acute attacks | at 3 months
  The number of asthma acute attacks refers to the total number of the patient's asthma acute attacks in the observation period after the completion of hydrogen treatment.
differentials from number of uses of first-aid drugs | at 3 months
  Number of uses of first aid drugs (short-term beta receptor stimulant) refers to the total number of administering salbutamol for relieving symptoms in the efficacy observation period after each subject completed hydrogen treatment.
differentials from Special allergens | at 3 months
  egg white, milk, fish, wheat, peanut, soybean (fx5); house dust, household dust mites, dust mites, cockroaches (hx2); Penicillium notatum/branch neurospora/Aspergillus fumigatus/Candida yeast/Alternaria neurospora/creep cinerea (mx2); inhaled allergen screening (Phadiatop); total IgE1.
differentials from blood routine examination | at 3 months
differentials from serum C reactive protein (CRP) | at 3 months
differentials from liver function examination | at 3 months
differentials from renal function examination | at 3 months
differentials from electrolyte test | at 3 months
differentials from routine urine test | at 3 months
differentials from 12-lead ECG test | at 3 months
differentials from urine pregnancy test for fertile women | at 3 months
differentials from pulmonary function | at 3 months
  Inspection items for patient pulmonary function include: FEV1.0, FEV1.0%, FVC, MMEF, MEF25, MEF50, MEF75, DLCO / VA, PEF †, FeNO, RV, TLC, RV / TLC, and FRC.
differentials from Baseline in Serum interleukin-6(IL-6) | at 3 months
differentials from Baseline in Serum interleukin-8( IL - 8) | at 3 months
differentials from Baseline in Serum tumor necrosis factor-a(TNF-a) | at 3 months
differentials from Baseline in Serum interleukin-4( IL - 4) | at 3 months
differentials from Baseline in Serum interleukin-5( IL - 5) | at 3 months
differentials from Baseline in Serum interleukin-13( IL - 13) | at 3 months
differentials from Baseline in Serum interleukin-17( IL - 17) | at 3 months
differentials from induced sputum test | at 3 months
  proportions of eosinophils, macrophages, lymphocytes, and neutrophils;

CONTACTS AND LOCATIONS:
Overall Officials: Nanshan Zhong, academician, Study Chair — China, Guangdong First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The main evaluation index and the secondary evaluation index of all participants will be share in 3 months after the end of this study.

REFERENCES:
- [Background] Sistek D, Tschopp JM, Schindler C, Brutsche M, Ackermann-Liebrich U, Perruchoud AP, Leuenberger P. Clinical diagnosis of current asthma: predictive value of respiratory symptoms in the SAPALDIA study. Swiss Study on Air Pollution and Lung Diseases in Adults. Eur Respir J. 2001 Feb;17(2):214-9. doi: 10.1183/09031936.01.17202140. PMID 11334122
- [Background] Holgate ST. Pathogenesis of asthma. Clin Exp Allergy. 2008 Jun;38(6):872-97. doi: 10.1111/j.1365-2222.2008.02971.x. PMID 18498538
- [Background] Sears MR. The definition and diagnosis of asthma. Allergy. 1993;48(17 Suppl):12-6; discussion 22-3. doi: 10.1111/j.1398-9995.1993.tb04692.x. PMID 8109702
- [Background] Hines SA. A Weekly Spark for Progressive Educators: Annie Murphy Paul's Brilliant Blog and Newsletter. J Microbiol Biol Educ. 2014 May 1;15(1):63-4. doi: 10.1128/jmbe.v15i1.716. eCollection 2014 May. No abstract available. PMID 24839527
- [Background] Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djukanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J. 2014 Feb;43(2):343-73. doi: 10.1183/09031936.00202013. Epub 2013 Dec 12. PMID 24337046
- [Background] Sly RM. Mortality from asthma. J Allergy Clin Immunol. 1989 Oct;84(4 Pt 1):421-34. doi: 10.1016/0091-6749(89)90351-5. No abstract available. PMID 2677091
- [Background] Bhavsar P, Hew M, Khorasani N, Torrego A, Barnes PJ, Adcock I, Chung KF. Relative corticosteroid insensitivity of alveolar macrophages in severe asthma compared with non-severe asthma. Thorax. 2008 Sep;63(9):784-90. doi: 10.1136/thx.2007.090027. Epub 2008 May 20. PMID 18492738
- [Background] Juniper EF, Guyatt GH, Ferrie PJ, Griffith LE. Measuring quality of life in asthma. Am Rev Respir Dis. 1993 Apr;147(4):832-8. doi: 10.1164/ajrccm/147.4.832. PMID 8466117
- [Background] Hew M, Bhavsar P, Torrego A, Meah S, Khorasani N, Barnes PJ, Adcock I, Chung KF. Relative corticosteroid insensitivity of peripheral blood mononuclear cells in severe asthma. Am J Respir Crit Care Med. 2006 Jul 15;174(2):134-41. doi: 10.1164/rccm.200512-1930OC. Epub 2006 Apr 13. PMID 16614347
- [Background] Wood LG, Gibson PG, Garg ML. Biomarkers of lipid peroxidation, airway inflammation and asthma. Eur Respir J. 2003 Jan;21(1):177-86. doi: 10.1183/09031936.03.00017003a. PMID 12570126
- [Background] Murata K, Fujimoto K, Kitaguchi Y, Horiuchi T, Kubo K, Honda T. Hydrogen peroxide content and pH of expired breath condensate from patients with asthma and COPD. COPD. 2014 Feb;11(1):81-7. doi: 10.3109/15412555.2013.830094. Epub 2013 Oct 10. PMID 24111595
- [Background] Montuschi P, Corradi M, Ciabattoni G, Nightingale J, Kharitonov SA, Barnes PJ. Increased 8-isoprostane, a marker of oxidative stress, in exhaled condensate of asthma patients. Am J Respir Crit Care Med. 1999 Jul;160(1):216-20. doi: 10.1164/ajrccm.160.1.9809140. PMID 10390403
- [Background] Zayasu K, Sekizawa K, Okinaga S, Yamaya M, Ohrui T, Sasaki H. Increased carbon monoxide in exhaled air of asthmatic patients. Am J Respir Crit Care Med. 1997 Oct;156(4 Pt 1):1140-3. doi: 10.1164/ajrccm.156.4.96-08056. PMID 9351613
- [Background] Wood LG, Garg ML, Simpson JL, Mori TA, Croft KD, Wark PA, Gibson PG. Induced sputum 8-isoprostane concentrations in inflammatory airway diseases. Am J Respir Crit Care Med. 2005 Mar 1;171(5):426-30. doi: 10.1164/rccm.200408-1010OC. Epub 2004 Dec 3. PMID 15579724
- [Background] Ohsawa I, Ishikawa M, Takahashi K, Watanabe M, Nishimaki K, Yamagata K, Katsura K, Katayama Y, Asoh S, Ohta S. Hydrogen acts as a therapeutic antioxidant by selectively reducing cytotoxic oxygen radicals. Nat Med. 2007 Jun;13(6):688-94. doi: 10.1038/nm1577. Epub 2007 May 7. PMID 17486089
- [Background] Kawamura T, Wakabayashi N, Shigemura N, Huang CS, Masutani K, Tanaka Y, Noda K, Peng X, Takahashi T, Billiar TR, Okumura M, Toyoda Y, Kensler TW, Nakao A. Hydrogen gas reduces hyperoxic lung injury via the Nrf2 pathway in vivo. Am J Physiol Lung Cell Mol Physiol. 2013 May 15;304(10):L646-56. doi: 10.1152/ajplung.00164.2012. Epub 2013 Mar 8. PMID 23475767
- [Background] Huang CS, Kawamura T, Peng X, Tochigi N, Shigemura N, Billiar TR, Nakao A, Toyoda Y. Hydrogen inhalation reduced epithelial apoptosis in ventilator-induced lung injury via a mechanism involving nuclear factor-kappa B activation. Biochem Biophys Res Commun. 2011 May 6;408(2):253-8. doi: 10.1016/j.bbrc.2011.04.008. Epub 2011 Apr 5. PMID 21473852
- [Background] Sun Q, Cai J, Liu S, Liu Y, Xu W, Tao H, Sun X. Hydrogen-rich saline provides protection against hyperoxic lung injury. J Surg Res. 2011 Jan;165(1):e43-9. doi: 10.1016/j.jss.2010.09.024. Epub 2010 Oct 15. PMID 21067781
- [Background] Zheng J, Liu K, Kang Z, Cai J, Liu W, Xu W, Li R, Tao H, Zhang JH, Sun X. Saturated hydrogen saline protects the lung against oxygen toxicity. Undersea Hyperb Med. 2010 May-Jun;37(3):185-92. PMID 20568549
- [Background] Terasaki Y, Ohsawa I, Terasaki M, Takahashi M, Kunugi S, Dedong K, Urushiyama H, Amenomori S, Kaneko-Togashi M, Kuwahara N, Ishikawa A, Kamimura N, Ohta S, Fukuda Y. Hydrogen therapy attenuates irradiation-induced lung damage by reducing oxidative stress. Am J Physiol Lung Cell Mol Physiol. 2011 Oct;301(4):L415-26. doi: 10.1152/ajplung.00008.2011. Epub 2011 Jul 15. PMID 21764987
- [Background] Ning Y, Shang Y, Huang H, Zhang J, Dong Y, Xu W, Li Q. Attenuation of cigarette smoke-induced airway mucus production by hydrogen-rich saline in rats. PLoS One. 2013 Dec 20;8(12):e83429. doi: 10.1371/journal.pone.0083429. eCollection 2013. PMID 24376700
- [Background] Xiao M, Zhu T, Wang T, Wen FQ. Hydrogen-rich saline reduces airway remodeling via inactivation of NF-kappaB in a murine model of asthma. Eur Rev Med Pharmacol Sci. 2013 Apr;17(8):1033-43. PMID 23661516
- [Background] Kajiyama S, Hasegawa G, Asano M, Hosoda H, Fukui M, Nakamura N, Kitawaki J, Imai S, Nakano K, Ohta M, Adachi T, Obayashi H, Yoshikawa T. Supplementation of hydrogen-rich water improves lipid and glucose metabolism in patients with type 2 diabetes or impaired glucose tolerance. Nutr Res. 2008 Mar;28(3):137-43. doi: 10.1016/j.nutres.2008.01.008. PMID 19083400
- [Background] Nakao A, Toyoda Y, Sharma P, Evans M, Guthrie N. Effectiveness of hydrogen rich water on antioxidant status of subjects with potential metabolic syndrome-an open label pilot study. J Clin Biochem Nutr. 2010 Mar;46(2):140-9. doi: 10.3164/jcbn.09-100. Epub 2010 Feb 24. PMID 20216947
- [Background] Kang KM, Kang YN, Choi IB, Gu Y, Kawamura T, Toyoda Y, Nakao A. Effects of drinking hydrogen-rich water on the quality of life of patients treated with radiotherapy for liver tumors. Med Gas Res. 2011 Jun 7;1(1):11. doi: 10.1186/2045-9912-1-11. PMID 22146004
- [Background] Ishibashi T, Sato B, Rikitake M, Seo T, Kurokawa R, Hara Y, Naritomi Y, Hara H, Nagao T. Consumption of water containing a high concentration of molecular hydrogen reduces oxidative stress and disease activity in patients with rheumatoid arthritis: an open-label pilot study. Med Gas Res. 2012 Oct 2;2(1):27. doi: 10.1186/2045-9912-2-27. PMID 23031079
- [Background] Ishibashi T, Sato B, Shibata S, Sakai T, Hara Y, Naritomi Y, Koyanagi S, Hara H, Nagao T. Therapeutic efficacy of infused molecular hydrogen in saline on rheumatoid arthritis: a randomized, double-blind, placebo-controlled pilot study. Int Immunopharmacol. 2014 Aug;21(2):468-73. doi: 10.1016/j.intimp.2014.06.001. Epub 2014 Jun 11. PMID 24929023